CLINICAL TRIAL: NCT03822442
Title: Cardiac MRI Increases Accuracy and Decreases Risk of Evaluation of Children with Cardiomyopathy and Cardiac Transplantation
Brief Title: MRI to Predict Rejection and Failure in Transplant and Cardiomyopathy Patients
Status: Recruiting | Type: Observational
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Laura Olivieri, Associate Professor of Pediatrics/Cardiologist, University of Pittsburgh
Other Study IDs: 11408
Record Dates: First submitted 2019-01-28; First posted 2019-01-30 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure; Cardiac Imaging Techniques; Congenital Heart Defects
Keywords: Cardiomyopathy, cardiomegaly; cardiac transplant
MeSH Terms: conditions — Heart Failure; Heart Defects, Congenital; Cardiomyopathies; Cardiomegaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Overall Research Strategy of this protocol is to refine and validate noninvasive CMR imaging sequences with invasive hemodynamic and pathology results to create a comprehensive, noninvasive, radiation-reduced regimen for pediatric cardiomyopathy and cardiac transplant assessment. We were the first to perform MR-guided cardiac catheterization in US children, and have accumulated the largest US experience, having performed over 75 procedures to date. Our unique experience puts us in strong position to leverage this technology to improve care of children with cardiomyopathy and transplant. Using an integrated approach, we will simultaneously (1) validate imaging measures of cardiac edema and fibrosis by correlating T1 and T2 map images with endomyocardial biopsy (EMB) results in Aim 1; (2) overlay T1, T2 map images into our x-ray system to display "hotspots" of T1 and T2 abnormalities to guide EMB in Aim 2; and (3) obtain radiation-free hemodynamic data in a highly vulnerable pediatric population by using CMR to guide catheter manipulation in the ICMR suite in Aim 3.

Age and diagnosis-matched historical controls will be identified from the last 10 years at Children's National as a control population for specific purposes of comparing (1) EMB yield without image overlay and (2) Radiation exposure during X-ray guided right heart catheterization. Identical information will be obtained and stored in the same 45CFR compliant database. Historical controls will be identified from the cardiac catheterization database by searching for age and diagnosis. A waiver of consent will be applicable here, as it would be inconvenient, insensitive and not feasible to consent families who have already undergone treatment.

DETAILED DESCRIPTION:
Anesthesia and Vascular Access After final review of protocol eligibility and of MRI safety, vascular access is obtained and sheaths are secured and covered with a sterile drape for transfer to the MRI. The catheterization is performed with continuous recording of electrocardiogram signals, transcutaneous hemoglobin ("pulse") oximetry, and under direct observation of an anesthesia licensed independent provider.

Diagnostic Cardiac MRI Before MRI catheterization begins, a focused cardiac MRI is performed to understand cardiac function and localize the proposed catheter trajectory from the access site into the targeted cardiovascular chambers.

MRI-guided catheterization Next during real-time MRI, a passive catheter is advanced from the access site into the targeted cardiovascular chambers under imaging guidance. Hemodynamic measurements (using fluid-filled transducers connected to the catheters) and blood hemoglobin saturation specimens are obtained from targeted cardiovascular chambers. Additional clinically-indicated and, if time allows, up to 30 minutes of research MRI is then performed before the subject is returned to the X-ray system.

Research MR Imaging Additional research cardiac MRI imaging to determine T1 and T2 values is undertaken next, with 6 short axis slices and one long axis slice positions identified for T1 map and T2 map acquisitions. The ICMR laboratory has a robust experience with acquisition of parametric mapping sequences. T1 and T2 maps will provide a roadmap for the cardiac biopsy that the patient requires in the xray suite.

Image Fusion to Guide Endomyocardial Biopsy At the conclusion of the MR imaging and MR-guided right heart catheterization procedure, the subject is returned to the X-ray suite for cardiac biopsy. Some cardiac biopsies are obtained in the usual fashion, and some biopsy specimens are obtained using image overlay software to display the regions of abnormal T1 and T2 onto the fluoroscopy system.

Conclusion of the procedure Following standard of care EMB, standard of care coronary angiography is obtained when if clinically indicated, all catheters and sheaths are removed and the subject is observed for complications in the cardiac procedure recovery unit or intensive care unit for at least 6 hours.

Diagnostic Echocardiogram Standard clinical data with strain analysis will be collected from the echocardiogram that is performed as a standard of care. Patients undergo a clinically indicated echocardiogram exam following the catheterization procedure in the Cardiac Post Recovery Unit (CPRU).

Blood Tests Serum for creatinine blood test will be collected at the time the clinically indicated IV is placed. Creatinine Is the standard test used at Children's National to assess kidney function. A total of 1cc of blood will be drawn to complete the test.

For subjects who consent to the optional study, an additional 5cc of blood work will be drawn at the time that the intravascular catheter is inserted for the clinically indicated cardiac catheterization procedure. The blood samples will be identified with the study ID number only, and will be stored in a secure freezer owned and maintained by the department of cardiology located at the Sheikh Zayed campus. This blood will be used to identify serum biomarkers, and to validate the potential use for diagnostic purposes.

Follow-up procedures At the conclusion of the procedure, the subject is returned to the X-ray table and all catheters are removed. The subject is observed for complications in an advanced nursing recovery unit or intensive care unit for at least 6 hours. The subject will be assessed for early and late complications at the time of discharge, and again approximately 2-6 weeks ± 7 days post procedure.

MRI Image Analysis In all cardiomyopathy and heart transplant patients, T1 measurements will be performed using offline analysis software according to our laboratory's measurement SOP for parametric maps. In heart transplant patients only, T2 measurements will be performed according to our laboratory's measurement SOP for parametric maps. Following measurements, images will be created for Image Overlay onto the fluoroscopy for patients undergoing clinically-indicated cardiac biopsy following the catheterization.

Biopsy Sample Analysis All biopsy samples will be evaluated clinically for evidence of cellular rejection, and a clinical report will be generated per clinical standard of care. In addition, each of the samples will undergo a separate staining procedure to identify regions of fibrosis. Digital images will be taken of the stained samples. Image processing software will be used to quantify percent fibrosis.

Historical Controls (for radiation exposure comparison, and biopsy yield comparison) Age and diagnosis-matched historical controls will be identified from the last 10 years at Children's National as a control population for specific purposes of comparing (1) EMB yield without image overlay and (2) Radiation exposure during X-ray guided right heart catheterization. Identical information will be obtained and stored in the same 45CFR compliant database. Historical controls will be identified from the cardiac catheterization database by searching for age and diagnosis. A waiver of consent will be applicable here, as it would be inconvenient, insensitive and not feasible to consent families who have already undergone treatment.

Subjects will not be provided additional information as a result of this research study.

Data will be reviewed in aggregate generating generalizable knowledge not applicable to an individual subject

ELIGIBILITY:
Inclusion Criteria:

* Children and adults of any age with heart transplant, suspected or confirmed cardiomyopathy
* Undergoing clinically-indicated ("medically necessary") cardiovascular catheterization

Exclusion Criteria:

* Cardiovascular instability including hemodynamic instability (such as requiring significant vasoactive infusion support) or mechanical hemodynamic support.
* Women who are pregnant
* Women who are nursing and who do not plan to discard breast milk for 24 hours
* Exclusion criteria for MRI

  * Central nervous system aneurysm clips
  * Implanted neural stimulator
  * Implanted cardiac pacemaker or defibrillator which are not MR safe or MR conditional according to the manufacturer
  * Cochlear implant
  * Ocular foreign body (e.g. metal shavings)
  * Implanted Insulin pump
  * Metal shrapnel or bullet.
* Exclusion criteria for Gadolinium

  * Renal disease with estimated glomerular filtration rate [eGFR] < 30 ml/min/1.73 m2 body surface area

The eGFR will be used to estimate renal function if reported by the laboratory.

The Schwartz equation 33 for estimation of GFR in children as recommended by the NKDEP is as follows:

GFR (mL/min/1.73 m2) = (k × height) / serum creatinine concentration

where k = constant defined as follows: k = 0.33 in premature infants k = 0.45 in term infants to 1 year of age k = 0.55 in children to 13 years of age k = 0.70 in adolescent males (not females because of the presumed increase in male muscle mass, the constant remains 0.55 for females) Height in cm Serum creatinine in mg/dL

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals referred to Children's National Medical Center with heart transplant or cardiomyopathy (i.e. "pre-transplant") to undergo clinically-indicated cardiac catheterization will be considered candidates for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlate MRI imaging results to biopsy results Correlate MRI imaging with endomyocardial biopsy | At the end of each catheterization procedure through study completion,up to 5 years
  Correlate MRI imaging sequences that can detect inflammation and fibrosis to quantities of inflammation and fibrosis seen on biopsy specimens taken from the same region.

SECONDARY OUTCOMES:
Compare yield of biopsy specimen collection using x-ray vs x-ray fused MRI images | At the end of each catheterization procedure through study completion,up to 5 years
  To compare the accuracy and yield of biopsy specimens collected for detection of rejection by using standard of care, unguided x-ray imaging for the biopsy to the accuracy and yield results of specimens collected using x-ray fused with MR imaging overlay for guidance towards "hotspots" of fibrosis and inflammation.
Radiation exposure | At the end of each catheterization procedure through study completion,up to 5 years
  To compare radiation exposure in this cohort of subjects (pre and post heart transplant) with recent historical controls undergoing matched invasive cardiology procedures at Children's National Medical Center prior to use of MR-guided cardiac catheterization.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Olivieri, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Health System, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Hsu DT, Pearson GD. Heart failure in children: part I: history, etiology, and pathophysiology. Circ Heart Fail. 2009 Jan;2(1):63-70. doi: 10.1161/CIRCHEARTFAILURE.108.820217. No abstract available. PMID 19808316
- [Background] Lee TM, Hsu DT, Kantor P, Towbin JA, Ware SM, Colan SD, Chung WK, Jefferies JL, Rossano JW, Castleberry CD, Addonizio LJ, Lal AK, Lamour JM, Miller EM, Thrush PT, Czachor JD, Razoky H, Hill A, Lipshultz SE. Pediatric Cardiomyopathies. Circ Res. 2017 Sep 15;121(7):855-873. doi: 10.1161/CIRCRESAHA.116.309386. PMID 28912187
- [Background] Lipshultz SE, Cochran TR, Briston DA, Brown SR, Sambatakos PJ, Miller TL, Carrillo AA, Corcia L, Sanchez JE, Diamond MB, Freundlich M, Harake D, Gayle T, Harmon WG, Rusconi PG, Sandhu SK, Wilkinson JD. Pediatric cardiomyopathies: causes, epidemiology, clinical course, preventive strategies and therapies. Future Cardiol. 2013 Nov;9(6):817-48. doi: 10.2217/fca.13.66. PMID 24180540
- [Background] McKenna WJ, Maron BJ, Thiene G. Classification, Epidemiology, and Global Burden of Cardiomyopathies. Circ Res. 2017 Sep 15;121(7):722-730. doi: 10.1161/CIRCRESAHA.117.309711. PMID 28912179
- [Background] Badano LP, Miglioranza MH, Edvardsen T, Colafranceschi AS, Muraru D, Bacal F, Nieman K, Zoppellaro G, Marcondes Braga FG, Binder T, Habib G, Lancellotti P; Document reviewers. European Association of Cardiovascular Imaging/Cardiovascular Imaging Department of the Brazilian Society of Cardiology recommendations for the use of cardiac imaging to assess and follow patients after heart transplantation. Eur Heart J Cardiovasc Imaging. 2015 Sep;16(9):919-48. doi: 10.1093/ehjci/jev139. Epub 2015 Jul 2. PMID 26139361
- [Background] Dayton JD, Kanter KR, Vincent RN, Mahle WT. Cost-effectiveness of pediatric heart transplantation. J Heart Lung Transplant. 2006 Apr;25(4):409-15. doi: 10.1016/j.healun.2005.11.443. Epub 2006 Feb 8. PMID 16563970
- [Background] Wagner K, Oliver MC, Boyle GJ, Miller SA, Law YM, Pigula F, Webber SA. Endomyocardial biopsy in pediatric heart transplant recipients: a useful exercise? (Analysis of 1,169 biopsies). Pediatr Transplant. 2000 Aug;4(3):186-92. doi: 10.1034/j.1399-3046.2000.00100.x. PMID 10933318
- [Background] Johnson JN, Hornik CP, Li JS, Benjamin DK Jr, Yoshizumi TT, Reiman RE, Frush DP, Hill KD. Cumulative radiation exposure and cancer risk estimation in children with heart disease. Circulation. 2014 Jul 8;130(2):161-7. doi: 10.1161/CIRCULATIONAHA.113.005425. Epub 2014 Jun 9. PMID 24914037
- [Background] Andreassi MG, Ait-Ali L, Botto N, Manfredi S, Mottola G, Picano E. Cardiac catheterization and long-term chromosomal damage in children with congenital heart disease. Eur Heart J. 2006 Nov;27(22):2703-8. doi: 10.1093/eurheartj/ehl014. Epub 2006 May 22. PMID 16717079
- [Background] Ait-Ali L, Andreassi MG, Foffa I, Spadoni I, Vano E, Picano E. Cumulative patient effective dose and acute radiation-induced chromosomal DNA damage in children with congenital heart disease. Heart. 2010 Feb;96(4):269-74. doi: 10.1136/hrt.2008.160309. Epub 2009 Aug 16. PMID 19687017
- [Background] Beels L, Bacher K, De Wolf D, Werbrouck J, Thierens H. gamma-H2AX foci as a biomarker for patient X-ray exposure in pediatric cardiac catheterization: are we underestimating radiation risks? Circulation. 2009 Nov 10;120(19):1903-9. doi: 10.1161/CIRCULATIONAHA.109.880385. Epub 2009 Oct 26. PMID 19858412
- [Background] Singh V, Mendirichaga R, Savani GT, Rodriguez A, Blumer V, Elmariah S, Inglessis-Azuaje I, Palacios I. Comparison of Utilization Trends, Indications, and Complications of Endomyocardial Biopsy in Native Versus Donor Hearts (from the Nationwide Inpatient Sample 2002 to 2014). Am J Cardiol. 2018 Feb 1;121(3):356-363. doi: 10.1016/j.amjcard.2017.10.021. Epub 2017 Oct 31. PMID 29197471
- [Background] Subherwal S, Kobashigawa JA, Cogert G, Patel J, Espejo M, Oeser B. Incidence of acute cellular rejection and non-cellular rejection in cardiac transplantation. Transplant Proc. 2004 Dec;36(10):3171-2. doi: 10.1016/j.transproceed.2004.10.048. PMID 15686721
- [Background] Parsai C, O'Hanlon R, Prasad SK, Mohiaddin RH. Diagnostic and prognostic value of cardiovascular magnetic resonance in non-ischaemic cardiomyopathies. J Cardiovasc Magn Reson. 2012 Aug 2;14(1):54. doi: 10.1186/1532-429X-14-54. PMID 22857649
- [Background] Piehler KM, Wong TC, Puntil KS, Zareba KM, Lin K, Harris DM, Deible CR, Lacomis JM, Czeyda-Pommersheim F, Cook SC, Kellman P, Schelbert EB. Free-breathing, motion-corrected late gadolinium enhancement is robust and extends risk stratification to vulnerable patients. Circ Cardiovasc Imaging. 2013 May 1;6(3):423-32. doi: 10.1161/CIRCIMAGING.112.000022. Epub 2013 Apr 18. PMID 23599309
- [Background] Olivieri L, Cross R, O'Brien KJ, Xue H, Kellman P, Hansen MS. Free-breathing motion-corrected late-gadolinium-enhancement imaging improves image quality in children. Pediatr Radiol. 2016 Jun;46(7):983-90. doi: 10.1007/s00247-016-3553-7. Epub 2016 Feb 17. PMID 26886912
- [Background] Kellman P, Arai AE. Cardiac imaging techniques for physicians: late enhancement. J Magn Reson Imaging. 2012 Sep;36(3):529-42. doi: 10.1002/jmri.23605. PMID 22903654
- [Background] Moon JC, Messroghli DR, Kellman P, Piechnik SK, Robson MD, Ugander M, Gatehouse PD, Arai AE, Friedrich MG, Neubauer S, Schulz-Menger J, Schelbert EB; Society for Cardiovascular Magnetic Resonance Imaging; Cardiovascular Magnetic Resonance Working Group of the European Society of Cardiology. Myocardial T1 mapping and extracellular volume quantification: a Society for Cardiovascular Magnetic Resonance (SCMR) and CMR Working Group of the European Society of Cardiology consensus statement. J Cardiovasc Magn Reson. 2013 Oct 14;15(1):92. doi: 10.1186/1532-429X-15-92. PMID 24124732
- [Background] Messroghli DR, Moon JC, Ferreira VM, Grosse-Wortmann L, He T, Kellman P, Mascherbauer J, Nezafat R, Salerno M, Schelbert EB, Taylor AJ, Thompson R, Ugander M, van Heeswijk RB, Friedrich MG. Clinical recommendations for cardiovascular magnetic resonance mapping of T1, T2, T2* and extracellular volume: A consensus statement by the Society for Cardiovascular Magnetic Resonance (SCMR) endorsed by the European Association for Cardiovascular Imaging (EACVI). J Cardiovasc Magn Reson. 2017 Oct 9;19(1):75. doi: 10.1186/s12968-017-0389-8. PMID 28992817
- [Background] Mavrogeni S, Bratis K, Georgakopoulos D, Karanasios E, Kolovou G, Pavlides G, Papadopoulos G. Evaluation of myocarditis in a pediatric population using cardiovascular magnetic resonance and endomyocardial biopsy. Int J Cardiol. 2012 Oct 18;160(3):192-5. doi: 10.1016/j.ijcard.2011.04.019. Epub 2011 May 10. PMID 21561672
- [Background] Kellman P, Wilson JR, Xue H, Ugander M, Arai AE. Extracellular volume fraction mapping in the myocardium, part 1: evaluation of an automated method. J Cardiovasc Magn Reson. 2012 Sep 10;14(1):63. doi: 10.1186/1532-429X-14-63. PMID 22963517
- [Background] Ugander M, Bagi PS, Oki AJ, Chen B, Hsu LY, Aletras AH, Shah S, Greiser A, Kellman P, Arai AE. Myocardial edema as detected by pre-contrast T1 and T2 CMR delineates area at risk associated with acute myocardial infarction. JACC Cardiovasc Imaging. 2012 Jun;5(6):596-603. doi: 10.1016/j.jcmg.2012.01.016. PMID 22698528
- [Background] Abu Hazeem AA, Dori Y, Whitehead KK, Harris MA, Fogel MA, Gillespie MJ, Rome JJ, Glatz AC. X-ray magnetic resonance fusion modality may reduce radiation exposure and contrast dose in diagnostic cardiac catheterization of congenital heart disease. Catheter Cardiovasc Interv. 2014 Nov 1;84(5):795-800. doi: 10.1002/ccd.25473. Epub 2014 Mar 20. PMID 24619541
- [Background] McGuirt D, Mazal J, Rogers T, Faranesh AZ, Schenke W, Stine A, Grant L, Lederman RJ. X-ray Fused With Magnetic Resonance Imaging to Guide Endomyocardial Biopsy of a Right Ventricular Mass. Radiol Technol. 2016 Jul;87(6):622-6. PMID 27390230
- [Background] Saikus CE, Lederman RJ. Interventional cardiovascular magnetic resonance imaging: a new opportunity for image-guided interventions. JACC Cardiovasc Imaging. 2009 Nov;2(11):1321-31. doi: 10.1016/j.jcmg.2009.09.002. PMID 19909937
- [Background] Ratnayaka K, Faranesh AZ, Hansen MS, Stine AM, Halabi M, Barbash IM, Schenke WH, Wright VJ, Grant LP, Kellman P, Kocaturk O, Lederman RJ. Real-time MRI-guided right heart catheterization in adults using passive catheters. Eur Heart J. 2013 Feb;34(5):380-9. doi: 10.1093/eurheartj/ehs189. Epub 2012 Aug 1. PMID 22855740